CLINICAL TRIAL: NCT06335888
Title: Cross-over, Randomized, Open-label, Single-centre, Phase II Clinical Trial to Investigate 18F-AzaFol in the Diagnosis of Large Vessel Vasculitis
Brief Title: A Clinical Trial to Investigate 18F-AzaFol in the Diagnosis of Large Vessel Vasculitis
Acronym: CRAFT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Paul Scherrer Institut, Center for Proton Therapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CRAFT
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Giant Cell Arteritis
Keywords: Tracer; PET imaging
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Intervention Model Description: Cross-over, randomized, open label, single-centre
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AzaFol first, FDG second (Experimental): AzaFol PET/CT imaging followed by FDG PET/CT imaging (standard of care)
  Interventions: Drug: AzaFol; Drug: FDG
- FDG first, AzaFol second (Active Comparator): FDG PET/CT imaging (standard of care) imaging followed by AzaFol PET/CT
  Interventions: Drug: AzaFol; Drug: FDG

INTERVENTIONS:
Drug: AzaFol — AzaFol-PET/CT imaging
Drug: FDG — FDG-PET/CT imaging

SUMMARY:
The goal of this open-label clinical trial is to evaluate the efficacy of AzaFol-PET/CT in the diagnosis of GCA (giant cell arteritis), to compare AzaFol- with 2-[18F]FDG-PET/CT, and to assess the safety and tolerability of AzaFol in subjects with suspicion of GCA.

Participants will undergo AzaFol-PET/CT imaging at a single timepoint.

DETAILED DESCRIPTION:
Giant cell arteritis (GCA) is the most common systemic vasculitis in the elderly population. 2-[18F]Fluor-2-desoxy-D-glucose (2-[18F]FDG) positron emission tomography (PET)/ computed tomography (CT) is performed to diagnose GCA (standard of care, SOC) but unable to reliably distinguish atherosclerosis from vasculitis. Activated macrophages express folate receptor (FR)-β and are enriched in inflamed vascular tissue in GCA. 3'-Aza-2'-[18F]Fluoro-Folic Acid (AzaFol) is a nuclear tracer targeting FRβ. The investigators hypothesize that AzaFol is a specific and reliable tracer to visualize activated macrophages in GCA and therefore might improve the discrimination of vasculitic and atherosclerotic lesions as compared to 2-[18F]FDG-PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 50 years with clinical suspicion of GCA
* Women of childbearing potential must not have a positive serum pregnancy test at the Screening Visit
* Subjects must be able to understand and adhere to all protocol requirements and must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.
* Are willing and able to comply with procedures required in this protocol.

Exclusion Criteria:

1. Folate deficiency
2. Female subjects who are pregnant, breastfeeding, or considering becoming pregnant during the study or within 30 days after the last dose of study drug
3. Concomitant treatment with medications that lead to a significant impairment of folic acid levels (methotrexate, pemetrexed, raltitrexed)
4. Concomitant glucose-containing infusion or parental nutrition within 6 hours prior to 2-[18F]FDG tracer application
5. Glucose level > 10 mmol/l at the timepoint of 2-[18F]FDG PET/CT
6. Unable to remain in the PET/CT for the duration of the examination
7. Unable to lie still for the duration of the examination (45 min)
8. Unable not to eat or drink (except water) for 6 hours prior to 2-[18F]FDG tracer application
9. Prior PET-imaging within 60 days before baseline
10. Intake of vitamin supplements containing > 1mg/day folic acid within 48 h prior to the PET/CT with AzaFol
11. Known hypersensitivity or allergy to folic acid
12. Enrolment of the investigator, his/her family members, employees and other dependent persons
13. Participation in another study with investigational drug within the 7 days preceding and during the present study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Specificity of the GCA-diagnosis at the patient level | Baseline
  Specificity of the GCA-diagnosis at the patient level using visual analysis as a diagnostic method with the clinical expert diagnosis as the reference standard

SECONDARY OUTCOMES:
Lesion detection rate (visual analysis) | Baseline
  Lesion detection rate in PET/CT in patients with suspicion of GCA, in patients with GCA (clinical expert diagnosis), and in patients without GCA (clinical expert diagnosis) by visual analysis at the level of the vessel.
Lesion detection rate (semiquantitative analysis) | Baseline
  Lesion detection rate in PET/CT in patients with suspicion of GCA, in patients with GCA (clinical expert diagnosis), and in patients without GCA (clinical expert diagnosis) by semiquantitative analysis at the level of the vessel.
Sensitivity of the GCA-diagnosis at the patient level | Baseline
  Sensitivity of the GCA-diagnosis at the patient level using visual evaluation as a diagnostic method with the clinical expert diagnosis as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Britta Maurer, Principal Investigator — Department of Rheumatology and Immunology, Inselspital, University of Bern, Bern, Switzerland
Locations (1):
- Department of Rheumatology and Immunology, University Hospital Bern, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No